CLINICAL TRIAL: NCT04236778
Title: A Phase 1a/1b, First-in-human, Open-label Study of Escalating Doses of VE303 in Healthy Adult Volunteers With or Without Vancomycin Pre-treatment to Evaluate Safety, Dosing, and Pharmacodynamics
Brief Title: First-in-human Study of VE303 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vedanta Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: VE303-01
Record Dates: First submitted 2020-01-09; First posted 2020-01-22 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Intervention Model Description: This Phase 1a/1b, first-in-human, open-label, single-center, dose-escalation study will evaluate the safety and microbiota changes induced by ingestion of VE303 following administration of oral vancomycin and VE303 administered without vancomycin pre-treatment in healthy adult subjects. Approximately 48 subjects are anticipated for enrollment, unless intermediate cohorts are required, in which case, up to an additional 18 subjects (for a total of approximately 66 subjects) may be enrolled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Cohort 1 (Experimental): Cohort 1 received oral vancomycin followed by a single dose of VE303.
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Cohort 2 (Experimental): Cohort 2 received oral vancomycin followed by a single day of 5 doses of VE303.
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Cohort 3 (Experimental): Cohort 3 received oral vancomycin followed by a single day of 10 doses of VE303.
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Cohort 4 (Experimental): Cohort 4 received oral vancomycin followed by 5 days of 10 doses daily of VE303.
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Cohort 5 (Experimental): Cohort 5 received oral vancomycin followed by 14 days of 10 capsules daily of VE303
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Cohort 6 (Experimental): Cohort 6 received 21 days of 10 doses daily of VE303
  Interventions: Drug: VE303
- Cohort 7 (Experimental): Cohort 7 received oral vancomycin followed by 10 doses of VE303 daily for 2 days, followed by 2 doses of VE303 daily for 3 days
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Cohort 8 (Experimental): Cohort 8 received oral vancomycin followed by 10 doses of VE303 daily for 2 days, followed by 2 doses of VE303 daily for 3 days
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Cohort 9 (Experimental): Cohort 8 received oral vancomycin followed by 10 doses of VE303 daily for 2 days, followed by 2 doses of VE303 daily for 3 days
  Interventions: Drug: VE303; Drug: Oral Vancomycin
- Vancomycin only (Placebo Comparator): This cohort only received oral vancomycin.
  Interventions: Drug: Oral Vancomycin

INTERVENTIONS:
Drug: VE303 — The VE303 Drug Product is a live biotherapeutic product (LBP) consisting of 8 clonal human commensal bacterial strains manufactured under GMP conditions.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 6; Cohort 7; Cohort 8; Cohort 9
Drug: Oral Vancomycin — Vancomycin, when taken by mouth, is used to treat Clostridium difficile-associated diarrhea.
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5; Cohort 7; Cohort 8; Cohort 9; Vancomycin only

SUMMARY:
This study was designed to evaluate safety and tolerability of a range of doses of VE303 in healthy adult volunteers. The study also evaluated pharmacokinetics of intestinal colonization by the VE303 strains and pharmacodynamics of recovery of the gut microbiota after administration of antibiotics followed by a course of VE303.

DETAILED DESCRIPTION:
VE303 is a rationally-defined bacterial consortium candidate being developed for the prevention of recurrent C. difficile infection. VE303 consists of 8 types of clonal human commensal bacteria strains selected for their ability to provide colonization resistance to C. difficile and manufactured under GMP conditions.

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who are judged to be in general good health
* Body mass index between 18.5 and 30 kg/m2
* Women either of non-child bearing potential or using a highly effective form of contraception
* Men using a highly effective method of contraception

Key Exclusion Criteria:

* Past or present clinically significant diseases that may affect the outcome of the study
* Taking any medications, herbal preparations, or natural substances, live bacteria products, or food that impacts or alter GI flora
* Use of proton pump inhibitors or other short or long acting antacid medications
* Taking or has received an investigation drug or treatment within 60 days of inpatient admission
* Known allergies to involved study drugs
* Chronic constipation or diarrhea
* History of or active IBD

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Safety of VE303 measured by incidence adverse events (AEs) | 12 months post-dose
  Measured in terms of incidence of AEs according to CTCAE V4.0
Tolerability of VE303 using modified PROMIS questionnaire (v1.0) | 12 months post-dose
  Characterized the highest well tolerated dose regimen of VE303 using modified PROMIS questionnaire (v1.0)

SECONDARY OUTCOMES:
Evaluate the colonization of the intestinal microbiota with VE303 component bacteria | 12 months post-dose
  Measurement of VE303 strain colonization in stool samples was performed using a metagenomic sequencing-based bioinformatic approach. A strain-specific marker panel was employed to characterize the relative abundance of VE303 strains in the intestinal microbiota.
Evaluate the changes in the intestinal microbiota due to VE303 dosing. | 12 months post-dose
  Measurement of intestinal microbiota due to VE303 dosing was performed using metagenomic sequencing- and metabolomic analysis-based approaches. Thus, focusing on taxonomic and functional changes occurring in the gut.
Evaluate the metabolomic changes in stool due to VE303 dosing. | 12 months post-dose
  Quantified changes in pool of metabolite levels (bile acids and short-chain fatty acids) from stool samples

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No